CLINICAL TRIAL: NCT04944186
Title: The Effect of Structured Pressure Injury Patient Education Program on Knowledge, Participation, Wound Healing Progress and Quality of Life Among Patient With Limited Mobility
Brief Title: Effect of Structured Pressure Injury Patient Education
Acronym: SPIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Deena @ Clare Thomas, Principal Investigator, University of Malaya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17033704
Record Dates: First submitted 2021-06-16; First posted 2021-06-29 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Pressure Injury; Limitation, Mobility
Keywords: patient education; structured patient education; wound healing; quality of life
MeSH Terms: conditions — Pressure Ulcer; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Prospective quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients in the experimental group will receive structured pressure injury patient education. It is consists of 2 sessions followed by biweekly follow-up for 8-week. The first session lasts for two days; the duration is 80 minutes (40 minutes /day for two days). Method of delivery is face to face, one to one with the aid of PowerPoint presentation and booklet. In the second session, the duration remains the same (80 minutes; 40 minutes/day for 2 days). The method of delivery also the same but teaching aid video presentation will be used. Three videos with a duration of approximately 2 - 3 minutes. In the second session, participants will be given a task to perform and document in the booklet given to monitoring its adherence. Upon completion of the two sessions, the patient will be follow-up biweekly and monitored their progress.
  Interventions: Other: Structured Pressure Injury Patient Education (mySPIPE)
- Control group (Other): Patients in this group shall continue with the standard patient education in the ward. Standard patient education routinely delivers through an informal verbal method after wound dressing is done.
  Interventions: Other: Standard Patient Education

INTERVENTIONS:
Other: Structured Pressure Injury Patient Education (mySPIPE) — It consists of PI education topics which include four main topics; 1) Pressure Injury: Why Me, which will be covering the basic information that patient need to know about PI; 2) Look After Your Skin, in this topics, patient will be thought about how skin checking was done and why it need to be done; 3) Preventing pressure injury, in this topic, patient will be emphasized on the suitable repositioning for them and the benefit of support surfaces and preventive wound dressing; 4) Help your PI heal, in this topic patient will be guided on what are condition that help PI healing and dietary needs to support wound healing
  Arms: Intervention Group
Other: Standard Patient Education — No fixed content/ duration of patient education. Basically, patient repositioning emphasized verbally after wound dressing completed.
  Arms: Control group

SUMMARY:
This study was planned as a prospective quasi-experimental study with the control group to determine the effect of structured pressure injury patient education (program on the knowledge, participation, wound healing progress, and quality of life among patients with limited mobility. We hypothesized that there would be a significant effect of structured pressure injury patient education on patient's knowledge, participation, wound healing rate, and quality of life between the control and intervention group over time.

DETAILED DESCRIPTION:
Patients with limited mobility and pressure injury are always at higher risk of having multiple functional, social, psychological, and financial repercussions. Without intensive PI management and prevention, these populations continue to suffer from prolonged pain, infection, social isolation, and exacerbation of mental health conditions.

While many preventive strategies and management are available to ease patient burden due to pressure injury, involving patient to take part in their care make a huge difference in patient outcome. In Malaysia, nurses play an important role in providing patient education on pressure injury, usually delivered through informal routine care, by distributing information leaflet or via digital resources on the Ministry of Health's website. However, the existing pressure injury education content is too broad, only emphasizing pressure injury prevention and no information on pressure injury care.

Few pieces of evidence reported on the effectiveness of patient education were able to improve patient knowledge on PI, increase patient participation in PI care associate with wound healing and improve the quality of life. However, there is a content gap in pressure injury patient education, which is wound care. While there a lot of patient education on pressure injury had been conducted extensively in the literature review, the components of wound care in pressure injury patient education are still unclear. Thus the primary objective of this study is to identify the effect of structured pressure injury patient education on the knowledge, participation, wound healing progress, and quality of life among patients with limited mobility. We hypothesized that there would be a significant effect of structured pressure injury patient education compared to the standard patient education on patient's knowledge, participation, wound healing rate, and quality of life between control and intervention group over time.

To achieve this research objective, we opt to conduct a quasi-experimental study-calculation of sample size is by using STATA 12.0 program. To calculate the sample size, power at 80%, and alpha was pre-set at 0.05. Mean, and standard deviation (σ) were extracted from previous researcher. Based on the calculation, a total of 120 eligible samples will be recruited with 60 samples each arm.

The patients included in the study will be assigned to the experimental group (structured pressure injury patient education) and control group (standard patient education). Eight medical-surgical wards including rehabilitation ward with a high prevalence of pressure injury were identified and invited to participate. Four wards agreed (medical ward, two multidisciplinary wards, and orthopedic ward), and the rest unable to participates because allocated as active COVID-19 ward. Thus, potential participants for this study will be recruited in these four wards in this tertiary hospital. The process of data collection will be started with control group first and followed by intervention group. Considering the limited availability of the target population set in the inclusion criteria earlier, the researcher opts to use convenience sampling.

For the implementation of the study, permission was obtained from the Medical Research Ethical Committee of the Malaysian Ministry of Health. The patient included in the study sample will be informed before the study that the study's purpose and participation are voluntary, and the patient may withdraw at any time without penalties.

Data collection tools; In this study, a checklist and structured questionnaires will be used to measure the four outcomes of this research which are 1) knowledge, 2) participation, 3) wound healing progress, and 4) quality of life.

Personal Information Checklist:

Checklists consist of three parts: part I- patient health status, part II: Wound Healing Progress (PUSH Tool 3.0), and part III- Nutritional Assessment (MNA-SF). This checklist will be filled up by the wound care nurse at baseline (T0), week-4 (T1), and week-8 (T2). The wound care nurse will be given a briefing and manual on how to fill-up the form. The wound care nurse responsible for filling up the required checklist is not aware of the study hypothesis.

Part I: Patient health status - patient's registration ID, gender, ward, IC number, age, comorbidities, PI categories, and PI site.

Part II: Wound Healing Progress (PUSH Tools 3.0) - to measure PI healing progress. The total score will be ranging between 0 to 17, lower PUSH tools 3.0 indicate better-wound healing progress.

Part II: Nutritional Status (MNA-SF) - to determine the patient's current nutritional status. It is further be classified into three categories: normal nutritional status (12-14 points), at risk of malnutrition (8-11 points), and malnourished (0 - 7 points). Measure once at baseline.

Questionnaires Part I: Sociodemographic - sociodemographic characteristics, including seven components: age, socio-economic status, gender, level of education level, ethnicity, occupation, and marital status.

Part II: Knowledge on Prevention and Treatment on Pressure Injury - use to self-assess basic knowledge of the prevention and treatment of pressure injury using Skin-Management Needs Assessment Checklist. The total score is expressed as a percentage and interpreted as a higher score reflecting better knowledge.

Part III: Patient Participation - self-administered questionnaire by which patient will self-rate their active participation based on the given items. The total score is expressed as a percentage and interpreted as a higher score reflecting greater participation.

Part IV: Quality of Life - PU-QOL questionnaire is a PI-specific questionnaire that measuring how much does the occurrence of PI bothers their life. Scale scores are generated by summing items and then transforming them to a 0-100 scale. High scores indicate more excellent patient bother.

Descriptive analysis The sociodemographic data of the patient will be described as frequencies and percentages for categorical data; mean and standard deviation for continuous data. Descriptive analysis was used to estimate the score of each outcome (patient's knowledge, participation, wound healing progress, and quality of life). The Chi-square test was used to test the crude associations for categorical data. Comparison between two groups of continuous variables will be made using an independent t-test. All analysis will be conducted at a 5% significant level.

Analysis of efficacy The effectiveness of the intervention will be assessed using repeated measure analysis of covariance (ANCOVA), modeling the within-subject effects. Model fit will be determined using residual plots and lack-of-fit tests. The effect sizes of the ANCOVA will be interpreted according to Cohen (a partial η2 of .01 can be considered a small effect, a partial η2 of .06 can be considered a medium effect, and a partial η2 of .14 can be considered a significant effect).

Potential risk, benefit, and patient's safety All potential participants will be ensured that patient safety will be the priority upon conducting this study. Participation in this study will not affect their treatment, and the risk is very minimal. They are free to decline to answer any of the questions that they feel uncomfortable with. The benefit of the study may vary, as reported in previous research. However, the information obtained from this study will help the patient to gain more understanding on pressure injury, how to prevent pressure injury in the future from getting worse, and knowledge on pressure injury care. A booklet on pressure injury education as education material will also be provided to patients in both control and intervention groups for future references.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be literate in either Malay or English language.
* Patients with PI stage II or stage III according to NPIAP staging of PI.
* PI located either at sacrococcygeal / greater trochanter/ischial tuberosities.
* Braden score 18 or less; with limited mobility
* Absence of any active malignant, hematological problem or psychiatric disease

Exclusion Criteria:

* Immunocompromised
* Having urinary/fecal incontinence
* Comatose patient or who are unable to respond verbally and cognitively impaired
* Patient who will undergo flap or skin graft surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Knowledge | 8 weeks
  Pressure Injury Knowledge (%)
Patient Participation | 8 weeks
  Patient Participation on Pressure Injury Prevention (%)
Wound-healing progress | 8 weeks
  Pressure injury condition includes size, exudate and tissue type (Score 0 -17). 0 minimum points indicate wound completely heal. Increasing number of score indicate wound condition is worsening. 17 maximum points represents a serious PI with wound area more than 24cm2 of of size, heavy exudate, and non-viable tissue.
Pressure ulcer-specific symptoms and functional outcomes | 8 weeks
  Pressure ulcer-specific symptoms and functional outcomes is assessed by the Pressure Ulcer Quality of Life (PU-QOL)

SECONDARY OUTCOMES:
Effectiveness of mySPIPE on PI knowledge | 8 weeks
  Effectiveness of mySPIPE on PI knowledge at week 4 and week 8. NAME OF MEASUREMENT : PI knowledge; MEASUREMENT TOOL - Questionnaire: Revised Skin-Management Needs Assessment Checklist (Revised SMNaC) ; UNIT OF MEASURE: Mean difference of PI knowledge at baseline (T0) to week 4 (T1), and Mean difference of PI knowledge from week 4 (T1) to week 8 (T2).
  Minimum value = 10, Maximum value = 100; Higher score better outcome.
Effectiveness of mySPIPE on Patient participation on PI prevention | 8 weeks
  Effectiveness of mySPIPE on patient participation on PI prevention at week 4 and week 8. NAME OF MEASUREMENT : Patient participation on PI prevention; MEASUREMENT TOOL - Questionnaire: Patient Participation on PI prevention (PPPIP); UNIT OF MEASURE: Mean difference of PPPIP at baseline (T0) to week 4 (T1), and Mean difference of PPPIP from week 4 (T1) to week 8(T2).
  Minimum value = 12.5, Maximum value = 100; Higher score better outcome.
Effectiveness of SPIPE on Wound Healing Progress | 8 weeks
  Effectiveness of SPIPE on Wound Healing Progress at week 4 and week 12. NAME OF MEASUREMENT : Wound Healing Progress; MEASUREMENT TOOL - Checklist : Pressure Ulcer Scale of Healing (PUSH 3.0); UNIT OF MEASURE: Mean difference of PUSH score at baseline (T0) to week 4 (T1), and Mean difference of PUSH score from week 4 (T1) to week 8 (T2).
  Minimum value = 0, Maximum value = 17; Lower score better outcome.
Effectiveness of mySPIPE on Pressure ulcer-specific symptoms and functional outcomes | 8 weeks
  Effectiveness of mySPIPE on Pressure ulcer-specific symptoms and functional outcomes at week 4 and week 8.
  NAME OF MEASUREMENT: Quality of Life; MEASUREMENT TOOL - Questionnaire: Pressure Ulcer Quality of Life (PUQOL); UNIT OF MEASURE: Mean difference of PUQOL at baseline (T0) to week 4 (T1), and Mean difference of PUQOL score from week 4 (T1) to week 8 (T2).
  Minimum value = 0, Maximum value = 100; Higher score better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Deena C Thomas, MNSc, Principal Investigator — University of Malaya; Chui Ping Lei, PhD, Study Director — University of Malaya; Abqariyah Yahya, PhD, Study Chair — University of Malaya; Alan Yap Jiann Wen, MSc; MD, Study Chair — Ministry of Health
Locations (1):
- Queen Elizabeth Hospital, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
IDP sharing plan include a study protocol, statistical analysis plan, and informed consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: October 2021 for 12 months
Access Criteria: Access granted upon request via direct email dnaclare@ums.edu.my

REFERENCES:
- [Background] Chaboyer W, Bucknall T, Webster J, McInnes E, Banks M, Wallis M, Gillespie BM, Whitty JA, Thalib L, Roberts S, Cullum N. INTroducing A Care bundle To prevent pressure injury (INTACT) in at-risk patients: A protocol for a cluster randomised trial. Int J Nurs Stud. 2015 Nov;52(11):1659-68. doi: 10.1016/j.ijnurstu.2015.04.018. Epub 2015 May 11. PMID 26003919
- [Background] Chaboyer W, Bucknall T, Webster J, McInnes E, Gillespie BM, Banks M, Whitty JA, Thalib L, Roberts S, Tallott M, Cullum N, Wallis M. The effect of a patient centred care bundle intervention on pressure ulcer incidence (INTACT): A cluster randomised trial. Int J Nurs Stud. 2016 Dec;64:63-71. doi: 10.1016/j.ijnurstu.2016.09.015. Epub 2016 Sep 23. PMID 27693836
- [Result] Robineau S, Nicolas B, Mathieu L, Durufle A, Leblong E, Fraudet B, Gelis A, Gallien P. Assessing the impact of a patient education programme on pressure ulcer prevention in patients with spinal cord injuries. J Tissue Viability. 2019 Nov;28(4):167-172. doi: 10.1016/j.jtv.2019.06.001. Epub 2019 Jun 22. PMID 31288977
- [Result] Kim JY, Cho E. Evaluation of a self-efficacy enhancement program to prevent pressure ulcers in patients with a spinal cord injury. Jpn J Nurs Sci. 2017 Jan;14(1):76-86. doi: 10.1111/jjns.12136. Epub 2016 Jul 7. PMID 28044436
- [Result] Arora M, Harvey LA, Glinsky JV, Chhabra HS, Hossain S, Arumugam N, Bedi PK, Lavrencic L, Hayes AJ, Cameron ID. Telephone-based management of pressure ulcers in people with spinal cord injury in low- and middle-income countries: a randomised controlled trial. Spinal Cord. 2017 Feb;55(2):141-147. doi: 10.1038/sc.2016.163. Epub 2016 Dec 20. PMID 27995939